CLINICAL TRIAL: NCT03297437
Title: Predictors for Successful Neurofeedback Training
Acronym: Predictors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frank Scharnowski (Other)
Responsible Party: Sponsor-Investigator, Frank Scharnowski, Prof. Dr., Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: PsychiatricUHZPUK
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neurofeedback training — In a neurofeedback setting, brain activity is measured non-invasively, the brain imaging data is analyzed in real-time, and then feedback regarding the current level of brain activity is provided to the subject.

SUMMARY:
The primary objective of this study is to identify predictors of neurofeedback training success.

DETAILED DESCRIPTION:
In the last decades, neurofeedback has been established as a promising scientific tool. Learning voluntary control over their own brain activity allows for establishing causal links between brain activity and mental functions. However, patients participants differ in their ability to learn control over their own brain activity with neurofeedback. It is thus crucial to understand why some participants are more successful in regulating their own brain activity than others. The objective of the present study is thus to identify predictors for successful learning self-regulation with real-time fMRI neurofeedback. To achieve this goal, we will evaluate the introspection ability of healthy participants using standardized psychological questionnaires and tasks. These scores will then be correlated with how well they learned self-regulation skills using established real-time fMRI neurofeedback protocols.

ELIGIBILITY:
Inclusion Criteria:

Age 18 - 65 years. Magnetic resonance imaging compatibility.

Exclusion Criteria:

Physical or psychiatric disorders (DSM-V diagnosis). Current substance abuse. Exclusion criteria applicable to MRI (metallic implants, claustrophobia, epilepsy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
correlation between introspection scores and learning success | 48 months
  The primary outcome measure is a correlation between introspection scores and neurofeedback learning success across all subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Psychiatry, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No